CLINICAL TRIAL: NCT02326337
Title: A Multi-national, Multi-center, Prospective, Randomized, Double Blinded, Placebo-controlled Trial to Evaluate the Efficacy of HyperBox Cyclical Topical Wound Oxygen Therapy (TWO2) in the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: Efficacy, Safety and Economic Benefits of Topical Wound Oxygen Therapy in the Treatment of Chronic Diabetic Foot Ulcers
Acronym: TWO2DFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AOTI Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOTI- TWO2DFU-01
Record Dates: First submitted 2014-11-19; First posted 2014-12-29 (Estimated); Results first posted 2025-04-20 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Group Sequential Design of a maximum of 220 subjects with two predetermined interim analyses at 73 and 146 subjects
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Topical Wound Oxygen Device (Active Comparator): Application of the Topical Wound Oxygen (TWO2) device that supplies cyclical oxygen pressure directly to the wound site within a sealed and humidified environment for 90 minutes, 5 times a week with Advanced Moist Wound Therapy (AMWT) dressings.
  Other Names:
  * Topical Wound Oxygen Therapy
  * TWO2
  Interventions: Device: TWO2 Device
- Placebo Device (Placebo Comparator): Application of placebo device that does not supply cyclical oxygen pressure directly to the wound site within a sealed and humidified environment for 90 minutes, 5 times a week with AMWT dressings.
  Interventions: Device: Placebo Device

INTERVENTIONS:
Device: TWO2 Device — Application of the Topical Wound Oxygen (TWO2) device that supplies cyclical oxygen pressure directly to the wound site within a sealed and humidified environment for 90 minutes, 5 times a week with AMWT dressings.
  Other Names: TWO2 Therapy
  Arms: Topical Wound Oxygen Device
Device: Placebo Device — Application of placebo device that does not supply cyclical oxygen pressure directly to the wound site within a sealed and humidified environment for 90 minutes, 5 times a week with AMWT dressings.
  Other Names: Sham Device, Control Device
  Arms: Placebo Device

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and economical benefits of Cyclical Pressure Topical Wound Oxygen (TWO2) Therapy in the treatment of chronic diabetic foot ulcers. Subjects will wear a standardized off-loading device and use advanced moist wound therapy (AMWT) dressings. Following a 2 week run-in period with the standardized care and after meeting all the eligibility criteria, half the subjects will use the TWO2 device, while the other half will use a sham device.

DETAILED DESCRIPTION:
Subjects meeting the initial eligibility criteria will enter a 2 week run-in period with a standardized off-loading device, advanced moist wound therapy (AMWT) dressings and will receive sharp debridement. Subjects with wounds that do not decrease more than 30% at the end of the 2 week run-in period and where all other eligibility criteria are met, will be randomized to either the TWO2 device arm, or sham (placebo) device arm.

All subjects will use the TWO2/Sham device for 90 minutes a day at their home or nursing care facility 5 times a week for the treatment phase of up to 12 weeks. Monitoring of the wound will take place with weekly clinic visits for safety and compliance assessment and documentation. Weekly wound photographs and measurements will be taken. Wounds that close at, or before, 12 weeks will continue to use TWO2/sham device, off-loading and AMWT and have an additional visit two weeks later to confirm wound closure. All subjects whether healed or not will enter a follow up period of an additional 12 and 38 weeks.

The maximum duration for participation in the trial is 54 weeks. During the follow-up phase, subjects will receive standard care according to the clinician's recommendation and will be asked not to participate in another wound care trial during this period.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a documented diagnosis of Diabetes mellitus Type 1 or 2
* Foot ulcer at or below ankle with duration of more than 4 weeks but no longer than 1 year
* If the index ulcer is a post amputation wound date of surgery must be > 30 days
* 2 week run in period with less than 30% wound size reduction
* University of Texas Grade 1A, 1B, 1C, 1D, 2A, 2B, 2C, or 2D (Appendix I)
* Ulcer is ≥ 1cm2 and ≤ 20cm2 after debridement at start of run-in period
* If more than one ulcer is present on the foot, only the largest is considered in the study (Index ulcer)
* Index ulcer must be ≥ 1cm away from any other ulcers present on the foot
* Adequate perfusion with ABI > 0.7 And TcpO2 > 30mmHg OR skin perfusion > 30mmHG OR Toe pressure > 30mmHg OR Duplex with biphasic waveforms below the knee
* No planned revascularization procedure or vascular surgery within the last/next 30 days
* Subject and/or caregiver are willing and able to comply with all specified care and visit requirements
* Subject has a reasonable expectation of completing the study; according to the Investigator's clinical judgment

Exclusion Criteria:

* Evidence of gangrene on any part of affected limb
* Documented evidence of osteomyelitis on any part of affected limb
* Index ulcer has exposed bone
* Index ulcer exhibits signs of severe clinical infection that requires hospitalization or immediate surgical intervention
* Active Charcot foot on the study limb
* Subject participated in another investigational device, drug or biological trial within last 30 days
* Uncontrolled diabetes: HbA1c > 12 %
* Renal dialysis or creatinine > 2.5
* Known immune insufficiency
* Chronic steroid use or immunosuppressive agents within the last three (3) months or is anticipated to require them during the course of the study
* Active treatment for malignancy (not specific to study limb)
* Patient has a Deep Vein Thrombosis within the last 30 days
* Subject has received growth factor therapy (e.g., autologous platelet-rich plasma gel, becaplermin, bilayered cell therapy, dermal substitute, extracellular matrix) within the screening period
* Subject may not be pregnant at the time of treatment

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Frykberg, DPM, Principal Investigator — Carl T. Hayden VA Medical Center
Locations (16):
- United States (9):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - NorthBay Center for Wounds, Vacaville, California
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - The Research Center Inc., Hialeah, Florida
  - Advanced Research Institute of Miami, Miami, Florida
  - Edward Hines, Jr. VA Hospital, Chicago, Illinois
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Salem VA Medical Center, Salem, Virginia
- France (3):
  - Avicenne Hospital, Bobigny
  - Hospital Simone Veil, Eaubonne
  - Montpellier University Hospital, Montpellier
- Städtisches Klinikum Dessau, Dessau, Germany
- Kirchberg Hospital, Luxembourg, Luxembourg
- United Kingdom (2):
  - Northwick Park Hospital, Harrow
  - King's College Hospital, London

REFERENCES:
- [Result] Frykberg RG, Franks PJ, Edmonds M, Brantley JN, Teot L, Wild T, Garoufalis MG, Lee AM, Thompson JA, Reach G, Dove CR, Lachgar K, Grotemeyer D, Renton SC; TWO2 Study Group. A Multinational, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Efficacy of Cyclical Topical Wound Oxygen (TWO2) Therapy in the Treatment of Chronic Diabetic Foot Ulcers: The TWO2 Study. Diabetes Care. 2020 Mar;43(3):616-624. doi: 10.2337/dc19-0476. Epub 2019 Oct 16. PMID 31619393

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Wound Oxygen Device: Application of the Topical Wound Oxygen (TWO2) device that supplies cyclical oxygen pressure directly to the wound site within a sealed and humidified environment for 90 minutes, 5 times a week with Advanced Moist Wound Therapy (AMWT) dressings.
  Other Names:
  * Topical Wound Oxygen Therapy
  * TWO2
  TWO2 Device: Application of the Topical Wound Oxygen (TWO2) device that supplies cyclical oxygen pressure directly to the wound site within a sealed and humidified environment for 90 minutes, 5 times a week with AMWT dressings.
Period: Overall Study
Arm/Group | Topical Wound Oxygen Device | Placebo Device
Started | 36 | 37
Completed | 36 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Wound Oxygen Device | Placebo Device | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (10.3) | 61.9 (9.5) | 63.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 32 | 31 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Hispanic | 26 | 24 | 50
  Black | 5 | 5 | 10
  Asian | 2 | 1 | 3
  American Indian | 0 | 1 | 1
  Not reported | 3 | 6 | 9
Diabetes Type 2 [Count of Participants; unit: Participants] | 32 | 33 | 65
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 30.8 (5.9) | 31.2 (7.6) | 31 (6.8)
Wound area (cm2) [Mean (Standard Deviation); unit: cm^2] | 3.02 (2.66) | 3.22 (2.54) | 3.13 (2.57)
Wound perimeter (cm) [Mean (Standard Deviation); unit: cm] | 6.22 (2.85) | 6.85 (4.18) | 6.54 (3.55)
Ulcer duration (days) [Mean (Standard Deviation); unit: Days] | 160.3 (96) | 174.6 (94) | 166.4 (95)
The University of Texas Staging System for Diabetic Foot Ulcers Grade I [Count of Participants; unit: Participants] — Grade IA: Superficial ulcer, not involving tendon capsule or bone Grade IB: With Infection Grade IC: With ischemia Grade ID: With infection and ischemia
  Participants | 22 | 31 | 53
The University of Texas Staging System for Diabetic Foot Ulcers Grade II [Count of Participants; unit: Participants] — Grade IIA: Ulcer penetrating to tendon or capsule Grade IIB: With Infection Grade IIC: With ischemia Grade IID: With infection and ischemia
  Participants | 14 | 6 | 20
Neuropathic foot [Count of Participants; unit: Participants] | 28 | 29 | 57
Smoker [Count of Participants; unit: Participants] | 13 | 10 | 23
Ankle brachial index, ratio (SD) [Mean (Standard Deviation); unit: Ratio] — The Ankle Brachial Index (ABI) is the systolic pressure at the ankle, divided by the systolic pressure at the arm. ABI has been shown to be a specific and sensitive metric for the diagnosis of Peripheral Arterial Disease (PAD).
  Normal ABI ranges from 1.0 - 1.4
  Values above 1.4 suggest a noncompressible calcified vessel.
  A value below 0.9 is considered diagnostic of PAD.
  Values less than 0.5 suggests severe PAD.
  (https://stanfordmedicine25.stanford.edu/the25/ankle-brachial-index.html)
  Ratio | 1.07 (0.23) | 1.00 (0.23) | 1.03 (0.23)
HbA1c, % (SD) [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] | 8.43 (1.75) | 8.14 (1.49) | 8.25 (1.64)

OUTCOME MEASURES:

1. Primary Outcome: Wound Closure Within 12 Weeks With the Use of Topical Wound Oxygen Therapy (TWO2)
Description: Number of Participants with complete wound closure defined as 100% skin re-epithelialization without dressing requirements which is confirmed by 2 consecutive study visits 2 weeks apart.
Time Frame: 12 weeks
Population: Patients with diabetic foot ulcers
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Wound Oxygen Device | Placebo Device
Number analyzed (Participants) | 36 | 37
Participants | 15 | 5

2. Secondary Outcome: Absolute Change in Ulcer Area
Description: Absolute change in ulcer area over 12 weeks in cm2
Time Frame: 12 weeks
Population: Patients with open ulcers
Measure: Mean (Standard Deviation); unit: cm2
Groups:
- Placebo: Application of placebo device that does not supply cyclical oxygen pressure directly to the wound site within a sealed and humidified environment for 90 minutes, 5 times a week with AMWT dressings.
  Placebo Device: Application of placebo device that does not supply cyclical oxygen pressure directly to the wound site within a sealed and humidified environment for 90 minutes, 5 times a week with AMWT dressings.
Arm/Group | Topical Wound Oxygen Device | Placebo
Number analyzed (Participants) | 36 | 37
cm2 | 1.97 (2.12) | .4 (0.041)

3. Secondary Outcome: Ulcer Recurrence
Description: Number of diabetic foot ulcers with recurrence at 12 months
Time Frame: 12 months
Population: Patient with closed diabetic foot ulcers
Measure: Number; unit: Count of wounds with recurrence
Arm/Group | Topical Wound Oxygen Device | Placebo Device
Number analyzed (Participants) | 15 | 5
Count of wounds with recurrence | 1 | 2

4. Secondary Outcome: Number of Amputation Events
Description: Number of amputation events during interventional period of the study.
Time Frame: 12 weeks
Population: Patients with Index limb amputations
Measure: Number; unit: Count of events
Arm/Group | Topical Wound Oxygen Device | Placebo Device
Number analyzed (Participants) | 36 | 37
Count of events | 2 | 3

5. Secondary Outcome: Incidence of Adverse Events
Description: Incidence of serious adverse events and adverse events
Time Frame: 54 weeks
Population: Patients with diabetic foot ulcers
Measure: Number; unit: Count of events
Arm/Group | Topical Wound Oxygen Device | Placebo Device
Number analyzed (Participants) | 36 | 37
Count of events
  Serious Adverse Events | 10 | 10
  Adverse Events | 8 | 8
  Device related death | 0 | 0

6. Secondary Outcome: Quality of Life Assessment
Description: The Cardiff Wound Impact Schedule questionnaire to measure quality of life. Measure of well-being items from each scale are summated, physical symptoms, everyday living and social life. The items are rated for the extent of the experience and each item is given a number value. This allows the patients to weight the items included in the scale. The well-being scale is scored on a 5-point Likert scale, with response options from 'strongly agree' to 'strongly disagree'. All three scales are then transformed onto a minimum = 0 up to a maximum = 100, where a low score indicates worse, and a high score indicates better feeling of well-being.
Time Frame: 12 weeks
Population: Study participants with open and healed ulcers.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Topical Wound Oxygen Device | Placebo Device
Number analyzed (Participants) | 36 | 37
units on a scale | 9.1 (13.9) | 0.1 (16.9)

7. Secondary Outcome: Economic Analysis
Description: Not performed or reported. Economic Analysis is a composite measure of the wound before the study (up to one year) and for the duration of the study. The assessment is obtained by documenting treatment history of the wound that includes types of dressings used, time taken for dressing changes, by whom dressings are changed, and type and duration of hospitalization as well as the administration of the EQ-5D questionnaire at the Baseline visit, weeks 4, 8 and 12 on treatment.
Time Frame: 12 weeks
Population: Patients with diabetic foot ulcers
Arm/Group | Topical Wound Oxygen Device | Placebo Device
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to Complete Wound Closure in Weeks
Description: Time to 100% wound closure utilizing Cox proportional hazards model, a statistical measure of difference of time to event (healing). Subjects who withdraw from treatment will be entered into the analysis and censored at the time they withdraw from the trial or are lost to follow up. The analysis will consider covariates that might influence the outcome in the trial.
Time Frame: 12 weeks or wound closure
Population: Time to complete wound closure, weeks.
Measure: Mean (Standard Deviation); unit: Weeks
Groups:
- Placebo: Application of placebo device that does not supply cyclical oxygen pressure directly to the wound site within a sealed and humidified environment for 90 minutes, 5 times a week with AMWT dressings.
Arm/Group | Topical Wound Oxygen Device | Placebo
Number analyzed (Participants) | 36 | 37
Weeks | 8.2 (1.9) | 6.3 (4.2)

ADVERSE EVENTS:
Time Frame: 54 Weeks (baseline up to maximum duration of study participation).
Description: Adverse Events were collected and assessed at every study visit by investigator.
Arm/Group | Topical Wound Oxygen Device | Placebo Device
All-Cause Mortality (participants affected / at risk) | 2/36 | 2/37
Serious Adverse Events (participants affected / at risk) | 6/36 | 7/37
Other Adverse Events (participants affected / at risk) | 6/36 | 7/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Wound Oxygen Device (N=36) | Placebo Device (N=37)
Wound Infection (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Hyperglycemic event (Endocrine disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Necrotic Tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cardiovascular Event (Cardiac disorders) | 1 (1) | 0 (0)
UTC Grade II Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Severe Maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Wound Oxygen Device (N=36) | Placebo Device (N=37)
UTC Grade I Ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Ulcer Decline (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Minor Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Minor Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Minor Necrotic Tissue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Edema (Vascular disorders) | 1 (1) | 1 (1)
Maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Deramatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Contusion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT02326337/Prot_SAP_000.pdf